CLINICAL TRIAL: NCT05369585
Title: An Open-label, Single Arm, Clinical Trial to Explore the Consumption Effects of TOTUM-63 on Metabolic Signatures, Microbiome, Energy Metabolism and Post-prandial Nutrient Processing in Individuals at Increased Cardio-metabolic Risk
Brief Title: Mode of Action (MoA) Study of TOTUM-63 in Individuals at Increased Cardio-metabolic Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Valbiotis (Industry)
Collaborators: Laval University (Other); Centre de Recherche de l'Institut Universitaire de Cardiologie et de Pneumologie de Quebec (Other); Valbiotis Canada inc. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2021-408; 255926 (Other: Health Canada); 2021-408 (Other: CERUL)
Record Dates: First submitted 2022-04-05; First posted 2022-05-11 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2022-05

CONDITIONS: Prediabetic State; Dysglycemia; Overweight and Obesity
Keywords: Dysglycemia; Prediabetes; Diabetes risk; Cardio-metabolic risk; Diet supplement; Plant extracts; Polyphenols; Microbiota; Magnetic Resonance Imaging
MeSH Terms: conditions — Prediabetic State; Overweight; Obesity | interventions — TOTUM-63

STUDY DESIGN:
Intervention Model Description: Open-label, single center, single arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TOTUM-63 (Experimental): Experimental active are supplemented with TOTUM-63, taken 3 times per day.
  Interventions: Dietary Supplement: TOTUM-63

INTERVENTIONS:
Dietary Supplement: TOTUM-63 — 5-g per day dose of TOTUM-63 supplement, a mix of 5 plant extracts. Daily dose for 8 weeks followed by a 4 weeks follow-up period without supplementation.

SUMMARY:
This clinical study aims to investigate the effects of TOTUM-63, a mix of 5 plant extracts, consumed at the daily regimen of three times per day, on cardiometabolic health and gut microbiota profile in overweight-obese individuals.

DETAILED DESCRIPTION:
In 2019, over 460 million adults had diabetes worldwide. Moreover, it was estimated by the International Diabetes Federation that about 700 million adults will have type 2 diabetes (T2D) by 2045. Valbiotis is a research & development company dedicated to scientific innovation for preventing and reducing the risk of metabolic and cardiovascular disease (CVD) using specific combinations of plant-based molecules. Valbiotis developed a formula (TOTUM-63) which is composed by the association of five plant extracts.

Given the results obtained in pre-clinical studies, as well as the good tolerance and first efficacy results of TOTUM-63 in two clinical trials on human subjects, this research aims to investigate the effects of TOTUM-63 on cardiometabolic health and gut microbiota profile in overweight-obese individuals. TOTUM-63 will be tested (5g acutely and 5g/d over 8 weeks of supplementation) on energy metabolism, post-prandial nutrients metabolism and hepatic health in overweight and obese subjects. Blood and feces samples collected before, and after the supplementation will allow to perform metabolomic, transcriptomic and metagenomics analyses to further explore the potential mechanisms of action of TOTUM-63.

ELIGIBILITY:
Main Inclusion Criteria:

* Body mass index (BMI) between ≥ 27 and < 40 kg/m2 kg/m²;
* Waist circumference > 94 cm for men and > 80 cm for women;
* Weight stable within ± 5% in the last three months;
* Fasting plasma TG ≥ 1.35 OR fasting glycemia ≥ 5.6 and ≤ 6.9 mmol/L OR HbA1c ≥ 5.6 and ≤ 6.4 %

Main Exclusion Criteria:

* Any metabolic disorder requiring pharmacological treatment and susceptible to affect glucose metabolism or plasma lipid levels or that might affect the study outcomes according to the investigator;
* Taking medication which may affect the study outcomes (or a medication modification less than 3 months prior to the study);
* To have taken regularly natural health products or enriched foods susceptible to modify the parameters followed by the investigator within the 3 months prior to the study;
* With a known or suspected food allergy, intolerance or hypersensitivity to any of the study products' ingredient as well as the non-medicinal ingredients of the product;
* Consuming more than 4 drinks of alcohol per week;
* Having a lifestyle deemed incompatible with the study according to the investigator including high level of physical activity (defined as more than 10 hours of intense physical activity a week, walking excluded);
* Pregnant or lactating women or intending to become pregnant within the timeframe of the study;
* Fasting blood triglycerides (TG) > 2.5 mmol/L;
* Fasting blood LDL-C > 4.9mmol/L or non-HDL-C > 5.7 mmol/L;
* Blood AST ≥ 45 U/L for men; and blood AST ≥ 35 U/L for women;
* Blood ALT ≥ 60 U/L for men; and blood ALT ≥ 50 U/L for women;
* Blood GGT ≥ 75 U/L for men; and blood GGT ≥ 50 U/L for women;
* Blood creatinine concentration > 125 μmol/L AND Estimated Glomerular Filtration Rate (eGFR) (calculated by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula) < 60 mL/min/1.73m²;
* Complete blood count (CBC) with hemoglobin < 120 g/L or leucocytes < 3000 /mm3 or leucocytes > 16000 /mm3 or clinically significant abnormality according to the investigator.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-04-25 (Actual); Primary Completion 2023-04-12 (Actual); Study Completion 2023-04-12 (Actual)

PRIMARY OUTCOMES:
Evolution of blood pressure | Baseline, V2 (4 weeks of intervention), V3 (8 weeks of intervention) and V4 (8 weeks of intervention + 4 weeks of follow-up)
  Systolic blood pressure, diastolic blood pressure (in mmHg)
Evolution of heart rate | Baseline, V2 (4 weeks of intervention), V3 (8 weeks of intervention) and V4 (8 weeks of intervention + 4 weeks of follow-up)
  Heart rate (in BPM)
Evolution of weight | Baseline, V2 (4 weeks of intervention), V3 (8 weeks of intervention) and V4 (8 weeks of intervention + 4 weeks of follow-up)
  Weight (in kg)
Evolution of waist circumference | Baseline, V2 (4 weeks of intervention), V3 (8 weeks of intervention) and V4 (8 weeks of intervention + 4 weeks of follow-up)
  Waist circumference (in cm)
Evolution of body mass index | Baseline, V2 (4 weeks of intervention), V3 (8 weeks of intervention) and V4 (8 weeks of intervention + 4 weeks of follow-up)
  Body mass index (in kg/m2)
Evolution of fasting glycemia | Baseline, V2 (4 weeks of intervention), V3 (8 weeks of intervention) and V4 (8 weeks of intervention + 4 weeks of follow-up)
  Fasting glycemia (in mmol/L)
Evolution of insulin secretion | Baseline, V2 (4 weeks of intervention), V3 (8 weeks of intervention) and V4 (8 weeks of intervention + 4 weeks of follow-up)
  Fasting insulinemia and C-peptide (in pmol/L)
Evolution of HbA1c | Baseline, V2 (4 weeks of intervention), V3 (8 weeks of intervention) and V4 (8 weeks of intervention + 4 weeks of follow-up)
  Fasting HbA1c (in %)
Evolution of satiety hormones | Baseline, V2 (4 weeks of intervention), V3 (8 weeks of intervention) and V4 (8 weeks of intervention + 4 weeks of follow-up)
  Peptide tyrosine tyrosine (PYY), cholecystokinin (in pg/ml)
Evolution of adipokines | Baseline, V2 (4 weeks of intervention), V3 (8 weeks of intervention) and V4 (8 weeks of intervention + 4 weeks of follow-up)
  Adiponectin, leptin, plasminogen activator inhibitor 1 (in ng/ml)
Evolution of inflammatory response (fibrinogen) | Baseline, V2 (4 weeks of intervention), V3 (8 weeks of intervention) and V4 (8 weeks of intervention + 4 weeks of follow-up)
  Fibrinogen (in ng/ml)
Evolution of inflammatory response (IL6, TNFa) | Baseline, V2 (4 weeks of intervention), V3 (8 weeks of intervention) and V4 (8 weeks of intervention + 4 weeks of follow-up)
  Interleukin 6, tumour necrosis factor alpha (in pg/ml)
Evolution of inflammatory response (hs-CRP) | Baseline, V2 (4 weeks of intervention), V3 (8 weeks of intervention) and V4 (8 weeks of intervention + 4 weeks of follow-up)
  High-sensitivity C-reactive protein (in mg/L)
Evolution of incretin response | Baseline, V2 (4 weeks of intervention), V3 (8 weeks of intervention) and V4 (8 weeks of intervention + 4 weeks of follow-up)
  Glucose-dependent insulinotropic polypeptide, glucagon-like peptide-1 (in pg/ml)
Evolution of blood lipid profile (lipid profile) | Baseline, V2 (4 weeks of intervention), V3 (8 weeks of intervention) and V4 (8 weeks of intervention + 4 weeks of follow-up)
  Triglycerides, total cholesterol, HDL-C, non-HDL-C, LDL-C, free-fatty-acids (in mmol/L)
Evolution of blood lipid profile (oxidized-LDL) | Baseline, V2 (4 weeks of intervention), V3 (8 weeks of intervention) and V4 (8 weeks of intervention + 4 weeks of follow-up)
  Oxidized-LDL (in ng/ml)
Evolution of blood lipid profile (ketones) | Baseline, V2 (4 weeks of intervention), V3 (8 weeks of intervention) and V4 (8 weeks of intervention + 4 weeks of follow-up)
  Ketones (in umol/L)
Evolution of fecal and plasma bile acid profiles | Baseline and V3 (8 weeks of intervention)
  Primary and secondary bile acids profiles (fecal and plasma) (in uM)
Evolution of metagenomic parameters (whole metagenome shotgun sequencing) | Baseline and V3 (8 weeks of intervention)
  Whole metagenome shotgun sequencing
Evolution of metagenomic parameters (microbiota diversity) | Baseline and V3 (8 weeks of intervention)
  Microbiota diversity measurements (Shannon index)
Evolution of metagenomic parameters (microbiota richness) | Baseline and V3 (8 weeks of intervention)
  Microbiota richness measurements (Simpson index)
Evolution of liver MRI | Baseline and V3 (8 weeks of intervention)
  Liver fat content
Evolution of FIB-4 index | Baseline, V2 (4 weeks of intervention), V3 (8 weeks of intervention) and V4 (8 weeks of intervention + 4 weeks of follow-up)
  FIB-4 index (FIB-4 index < 1.45 in the context of steatosis allows the exclusion of a clinically significant fibrosis)
Evolution of BARD score | Baseline, V2 (4 weeks of intervention), V3 (8 weeks of intervention) and V4 (8 weeks of intervention + 4 weeks of follow-up)
  BARD score (from 0 to 4, with a score of 4 resulting in a higher risk of advanced fibrosis)
Evolution of NAFLD fibrosis score | Baseline, V2 (4 weeks of intervention), V3 (8 weeks of intervention) and V4 (8 weeks of intervention + 4 weeks of follow-up)
  NAFLD fibrosis score (< -1.455 low fibrosis probability; -1.455 to 0.676 intermediate score; > 0.676 high probability of fibrosis)
Evolution in kinetics of glucose metabolism | Baseline, V2 (4 weeks of intervention), V3 (8 weeks of intervention) and V4 (8 weeks of intervention + 4 weeks of follow-up)
  Evaluation of glucose concentrations during a 6-hours mixed-meal tolerance test (in mmol/L)
Evolution in kinetics of insulin secretion | Baseline, V2 (4 weeks of intervention), V3 (8 weeks of intervention) and V4 (8 weeks of intervention + 4 weeks of follow-up)
  Evaluation of blood insulin and C-peptide during a 6-hours mixed-meal tolerance test (in pmol/L)
Evolution in kinetics of blood lipid profile | Baseline, V2 (4 weeks of intervention), V3 (8 weeks of intervention) and V4 (8 weeks of intervention + 4 weeks of follow-up)
  Evaluation of triglycerides, total cholesterol, HDL-C, non-HDL-C and LDL-C during a 6-hours mixed-meal tolerance test (in mmol/L)
Evolution of kinetics of incretin parameters | Baseline, V2 (4 weeks of intervention), V3 (8 weeks of intervention) and V4 (8 weeks of intervention + 4 weeks of follow-up)
  Evaluation of glucose-dependent insulinotropic polypeptide, glucagon-like peptide-1 during a 2-hours mixed-meal tolerance test (in pg/ml)
Evolution of inflammatory parameters (fibrinogen) | Baseline, V2 (4 weeks of intervention), V3 (8 weeks of intervention) and V4 (8 weeks of intervention + 4 weeks of follow-up)
  Evaluation of fibrinogen before and after a 6-hours mixed-meal tolerance test (in ng/ml)
Evolution of inflammatory parameters (IL6, TNFA) | Baseline, V2 (4 weeks of intervention), V3 (8 weeks of intervention) and V4 (8 weeks of intervention + 4 weeks of follow-up)
  Evaluation of interleukin 6, tumour necrosis factor alpha before and after a 6-hours mixed-meal tolerance test (in pg/ml)
Evolution of inflammatory parameters (hs-CRP) | Baseline, V2 (4 weeks of intervention), V3 (8 weeks of intervention) and V4 (8 weeks of intervention + 4 weeks of follow-up)
  Evaluation high-sensitivity C-reactive protein before and after a 6-hours mixed-meal tolerance test (in mg/L)
Evolution of energy metabolism (respiratory quotient) | Baseline, V2 (4 weeks of intervention), V3 (8 weeks of intervention) and V4 (8 weeks of intervention + 4 weeks of follow-up)
  Evaluation of respiratory quotient before and after a 6-hours mixed-meal tolerance test (in carbon dioxide (CO2) eliminated / dioxygen (O2) consumed)
Evolution of energy metabolism (resting metabolic rate) | Baseline, V2 (4 weeks of intervention), V3 (8 weeks of intervention) and V4 (8 weeks of intervention + 4 weeks of follow-up)
  Evaluation of resting metabolic rate before and after a 6-hours mixed-meal tolerance test (in kcal/day)
Evolution of energy metabolism (energy expenditure) | Baseline, V2 (4 weeks of intervention), V3 (8 weeks of intervention) and V4 (8 weeks of intervention + 4 weeks of follow-up)
  Evaluation of energy expenditure before and after a 6-hours mixed-meal tolerance test (in kcal/kg/h)

SECONDARY OUTCOMES:
Evolution of Safety parameters (hepatic enzymes) | Baseline, V2 (4 weeks of intervention), V3 (8 weeks of intervention) and V4 (8 weeks of intervention + 4 weeks of follow-up)
  Aspartate aminotransferase (AST), alanine aminotransferase (ALT), gamma-glutamyltransferase (GGT) (in U/L)
Evolution of Safety parameters (AST/ALT ratio) | Baseline, V2 (4 weeks of intervention), V3 (8 weeks of intervention) and V4 (8 weeks of intervention + 4 weeks of follow-up)
  AST/ALT ratio
Evolution of Safety parameters (albumin) | Baseline, V2 (4 weeks of intervention), V3 (8 weeks of intervention) and V4 (8 weeks of intervention + 4 weeks of follow-up)
  Albumin (in g/L)
Evolution of Safety parameters (creatinine) | Baseline, V2 (4 weeks of intervention), V3 (8 weeks of intervention) and V4 (8 weeks of intervention + 4 weeks of follow-up)
  Creatinine (in umol/L)
Evolution of complete blood count (red and white blood cells, platelet) | Baseline, V2 (4 weeks of intervention), V3 (8 weeks of intervention) and V4 (8 weeks of intervention + 4 weeks of follow-up)
  Red blood cells, white blood cells, platelet (in cells/mm3)
Evolution of complete blood count (hemoglobin) | Baseline, V2 (4 weeks of intervention), V3 (8 weeks of intervention) and V4 (8 weeks of intervention + 4 weeks of follow-up)
  Hemoglobin (in g/L)
Evolution of complete blood count (hematocrit) | Baseline, V2 (4 weeks of intervention), V3 (8 weeks of intervention) and V4 (8 weeks of intervention + 4 weeks of follow-up)
  Hematocrit (in %)
Evolution of transcriptomics | Baseline and V3 (8 weeks of intervention)
  RNA sequencing
Evolution of metabolomics (amino acids, fatty acids and acylcarnitine species) | Baseline and V3 (8 weeks of intervention)
  Evolution of amino acids, fatty acids and acylcarnitine species (in uM)

CONTACTS AND LOCATIONS:
Overall Officials: André Marette, PhD, Principal Investigator — Laval University; Patrick Couture, MD FRCP PhD, Principal Investigator — Laval University
Locations (1):
- Institute of Nutrition and Funtional Foods (INAF) - Laval University, Québec, Canada

IPD SHARING:
Plan to Share IPD: No